CLINICAL TRIAL: NCT03598985
Title: Validity and Reliability of a Smartphone Application for Assessing Balance in Patients With Chronic Ankle Instability
Brief Title: Smartphone for Assessing Balance in Patients With Ankle Instability
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aliaa Rehan Youssef, assistant professor, Cairo University
Other Study IDs: NAbdo
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Chronic Ankle Instability
Keywords: Balance; Smartphone; Validity; Reliability; chronic ankle instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CAI: Patients referred with a confirmed diagnosis of CAI, with a Cumberland Ankle Instability tool score lower than 27 points. Patients should have had a recurrent sprain within the previous year.
  Patients will have their balance assessed using the "Myankle" smartphone application simultaneously with Biodex balance system assessment.
  Interventions: Diagnostic Test: Smartphone "MyAnkle" balance application
- Healthy participants: Healthy participants who are not complaining of pain and have not be exposed to trauma, injury or undergone surgery for the lower quadrant of the body.
  Participants will have their balance assessed using the "MyAnkle" smartphone application simultaneously with Biodex balance system assessment.
  Interventions: Diagnostic Test: Smartphone "MyAnkle" balance application

INTERVENTIONS:
Diagnostic Test: Smartphone "MyAnkle" balance application — Balance will be assessed simultaneously using "MyAnkle" application and the Biodex balance system. The smartphone will be fixed to the middle of the shin with an armband. Participants will assume a single leg stance on each side under two conditions: eyes opened and closed. Testing will be done at three levels of difficulty; least difficult (level 8), moderate (level 6) and severe difficult (level 4). A conditioning trial for each level will be given for 30 seconds. Further, a 2-minute rest between tests will be given. During the testing, participants should not touch the ground or stance limb by other limb nor to grasp the handrail. Participants will repeat the same testing in two separate sessions, with one-week interval in between.
  Other Names: Biodex Balance system

SUMMARY:
This study aims at investigating the validity and reliability of a smartphone application "MyAnkle: in assessing the balance component of postural control in patients with chronic ankle instability (CAI).

DETAILED DESCRIPTION:
Lateral ankle sprain (LAS) is a common injury in athletic and regular activities; with an incidence of 7 per 1000 exposure. After LAS, residual symptoms may persist leading to chronic ankle instability (CAI). This instability is believed to arise from dysfunctional postural control, defective proprioception, weak muscles, or reduced ankle range of motion (ROM).Thus, assessment of postural control is essential for proper clinical decision-making and treatment selection.

With advances in technology, smartphone has been introduced as an assessment tool for the musculoskeletal system. For example, it was used in assessment of ROM and mobility in stroke patients and frail elderly conditions. Further, it was used to assess balance and falling risk in those population. In addition, it was used to assess balance in healthy and participants with chronic ankle sprain. These studies proved that smartphone is a valid and reliable tool that is light in weight and inexpensive. Yet, these studies have some methodological concerns. For example, the application was not validated against gold standard or was validated only in healthy volunteers rather than in patients with musculoskeletal dysfunction. Further, a few of these studies did not establish the application discriminative validity between patients and healthy controls. Thus, this study will try to answer the following question: "Is smartphone application a valid and reliable tool to assess balance in patients with CAI compared to gold standards?

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aging from 18 to 35 years old.
2. Referred with a confirmed diagnosis of CAI, with a Cumberland Ankle Instability tool score lower than 27 points.
3. Had a recurrent sprain within the previous year.

Exclusion Criteria:

1. History of major surgery of lower limb or spine.
2. History of ankle fracture or any other lower limb fracture in the past 2 years.
3. History of lower limb injury 3 months prior to study.
4. Presence of problems that affect balance performance as visual or vestibular deficits, neurologic disease, or cerebral concussions during the past 3 months.
5. Being currently enrolled in a balance training rehabilitation program.
6. Weakness of lower limb musculatures or trunk upon screening muscle testing by the investigator.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifty patients with CAI and 50 gender-, BMI and age-matched healthy volunteers will be enrolled in this study.
  Healthy participants will be recruited from undergraduate and graduate students of the faculty of Physical Therapy, Cairo University, Egypt. All healthy subjects will be asymptomatic with no neuromusculoskeletal signs or symptoms.
  Male and female adult patients with CAI will be recruited from the outpatient clinic of the faculties of Physical Therapy and Medicine, Cairo University, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Concurrent validity of smartphone MyAnkle application | One day
  Correlation between the score of "MyAnkle" smartphone balance application and stability score of the Biodex balance system.

SECONDARY OUTCOMES:
Intrarater reliability of smartphone measurements | one week
  same investigator will repeat balance assessment using "MyAnkle" smartphone balance application
Interrater reliability of smartphone measurements | one day
  Three investigators will assess balance using the MyAnkle smartphone application

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Rehan Youssef, PhD, Principal Investigator — Cairo University, Faculty of Physical Therapy
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Anandacoomarasamy A, Barnsley L. Long term outcomes of inversion ankle injuries. Br J Sports Med. 2005 Mar;39(3):e14; discussion e14. doi: 10.1136/bjsm.2004.011676. PMID 15728682
- [Background] Bahr R, Karlsen R, Lian O, Ovrebo RV. Incidence and mechanisms of acute ankle inversion injuries in volleyball. A retrospective cohort study. Am J Sports Med. 1994 Sep-Oct;22(5):595-600. doi: 10.1177/036354659402200505. PMID 7810781
- [Background] Capela NA, Lemaire ED, Baddour N, Rudolf M, Goljar N, Burger H. Evaluation of a smartphone human activity recognition application with able-bodied and stroke participants. J Neuroeng Rehabil. 2016 Jan 20;13:5. doi: 10.1186/s12984-016-0114-0. PMID 26792670
- [Background] Chiu YL, Tsai YJ, Lin CH, Hou YR, Sung WH. Evaluation of a smartphone-based assessment system in subjects with chronic ankle instability. Comput Methods Programs Biomed. 2017 Feb;139:191-195. doi: 10.1016/j.cmpb.2016.11.005. Epub 2016 Nov 11. PMID 28187890
- [Background] Delahunt E, Monaghan K, Caulfield B. Changes in lower limb kinematics, kinetics, and muscle activity in subjects with functional instability of the ankle joint during a single leg drop jump. J Orthop Res. 2006 Oct;24(10):1991-2000. doi: 10.1002/jor.20235. PMID 16894592
- [Background] Delahunt E, Monaghan K, Caulfield B. Altered neuromuscular control and ankle joint kinematics during walking in subjects with functional instability of the ankle joint. Am J Sports Med. 2006 Dec;34(12):1970-6. doi: 10.1177/0363546506290989. Epub 2006 Aug 22. PMID 16926342
- [Background] Doherty C, Delahunt E, Caulfield B, Hertel J, Ryan J, Bleakley C. The incidence and prevalence of ankle sprain injury: a systematic review and meta-analysis of prospective epidemiological studies. Sports Med. 2014 Jan;44(1):123-40. doi: 10.1007/s40279-013-0102-5. PMID 24105612
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Background] Freeman MA, Dean MR, Hanham IW. The etiology and prevention of functional instability of the foot. J Bone Joint Surg Br. 1965 Nov;47(4):678-85. No abstract available. PMID 5846767
- [Background] Garrick JG. The frequency of injury, mechanism of injury, and epidemiology of ankle sprains. Am J Sports Med. 1977 Nov-Dec;5(6):241-2. doi: 10.1177/036354657700500606. No abstract available. PMID 563179
- [Background] Patterson JA, Amick RZ, Thummar T, Rogers ME. Validation of measures from the smartphone sway balance application: a pilot study. Int J Sports Phys Ther. 2014 Apr;9(2):135-9. PMID 24790774
- [Background] Triantafyllidis AK, Velardo C, Salvi D, Shah SA, Koutkias VG, Tarassenko L. A Survey of Mobile Phone Sensing, Self-Reporting, and Social Sharing for Pervasive Healthcare. IEEE J Biomed Health Inform. 2017 Jan;21(1):218-227. doi: 10.1109/JBHI.2015.2483902. Epub 2015 Sep 29. PMID 26441432
- [Background] Mourcou Q, Fleury A, Diot B, Vuillerme N. iProprio: a smartphone-based system to measure and improve proprioceptive function. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:2622-2625. doi: 10.1109/EMBC.2016.7591268. PMID 28268860
- [Background] Perron M, Hebert LJ, McFadyen BJ, Belzile S, Regniere M. The ability of the Biodex Stability System to distinguish level of function in subjects with a second-degree ankle sprain. Clin Rehabil. 2007 Jan;21(1):73-81. doi: 10.1177/0269215506071288. PMID 17213244
- [Background] Roeing KL, Hsieh KL, Sosnoff JJ. A systematic review of balance and fall risk assessments with mobile phone technology. Arch Gerontol Geriatr. 2017 Nov;73:222-226. doi: 10.1016/j.archger.2017.08.002. Epub 2017 Aug 4. PMID 28843965
- [Background] Ross SE, Guskiewicz KM. Examination of static and dynamic postural stability in individuals with functionally stable and unstable ankles. Clin J Sport Med. 2004 Nov;14(6):332-8. doi: 10.1097/00042752-200411000-00002. PMID 15523204
- [Background] Hertel J. Functional Anatomy, Pathomechanics, and Pathophysiology of Lateral Ankle Instability. J Athl Train. 2002 Dec;37(4):364-375. PMID 12937557
- [Background] Ross SE, Guskiewicz KM, Gross MT, Yu B. Balance measures for discriminating between functionally unstable and stable ankles. Med Sci Sports Exerc. 2009 Feb;41(2):399-407. doi: 10.1249/MSS.0b013e3181872d89. PMID 19127184
- [Background] Schwenk M, Mohler J, Wendel C, D'Huyvetter K, Fain M, Taylor-Piliae R, Najafi B. Wearable sensor-based in-home assessment of gait, balance, and physical activity for discrimination of frailty status: baseline results of the Arizona frailty cohort study. Gerontology. 2015;61(3):258-67. doi: 10.1159/000369095. Epub 2014 Dec 24. PMID 25547185
- [Background] Shah N, Aleong R, So I. Novel Use of a Smartphone to Measure Standing Balance. JMIR Rehabil Assist Technol. 2016 Mar 29;3(1):e4. doi: 10.2196/rehab.4511. PMID 28582247
- [Background] Testerman C, Vander Griend R. Evaluation of ankle instability using the Biodex Stability System. Foot Ankle Int. 1999 May;20(5):317-21. doi: 10.1177/107110079902000510. PMID 10353771